CLINICAL TRIAL: NCT01497938
Title: ASPIRE (Automation to Simulate Pancreatic Insulin Response): Pivotal In Home Study to Determine Safety and Efficacy of the LGS Feature in Sensor-augmented Pumps
Brief Title: Outpatient Study to Evaluate Safety and Effectiveness of the Low Glucose Suspend Feature
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 237
Record Dates: First submitted 2011-12-18; First posted 2011-12-23 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Glucose Suspend feature (LGS) (Experimental): According to randomization, Low Glucose Suspend (LGS) will be turned ON in the treatment arm of the study
  Interventions: Device: Medtronic MMT-754 Veo Insulin pump testing Low Glucose Suspend (LGS) feature
- Control Arm (Experimental): The Low Glucose Suspend feature will not be available to subjects in the control arm
  Interventions: Device: Medtronic (NO LGS FEATURE ) using Paradigm® Revel™2.0 Pump

INTERVENTIONS:
Device: Medtronic MMT-754 Veo Insulin pump testing Low Glucose Suspend (LGS) feature — Automatic suspension of insulin delivery when glucose is low.
  Arms: Low Glucose Suspend feature (LGS)
Device: Medtronic (NO LGS FEATURE ) using Paradigm® Revel™2.0 Pump — No Automatic suspension of insulin delivery when glucose is low.
  Arms: Control Arm

SUMMARY:
Introduction:

The purpose of the pivotal In Home study is to collect clinical data on the safety and efficacy of the Paradigm LGS System in the actual use environment and by the intended use population. ASPIRE is a multi-center, in home, randomized parallel adaptive study design with type 1 diabetes. The study will compare A1C and CGM based nocturnal hypoglycemic events in a treatment arm to a control arm. Arms are defined as:

* Treatment Arm (LGS ON) using Paradigm® VEO™ Pump
* Control Arm (NO LGS FEATURE ) using Paradigm® Revel™2.0 Pump

The study's objectives are two-fold:

1. The first study objective is to demonstrate that home use of Low Glucose Suspend (LGS) is safe and is not associated with glycemic deterioration, as measured by change in A1C from baseline to end of study participation.
2. The second study objective is to demonstrate that home use of Low Glucose Suspend (LGS) is associated with reduction in nocturnal hypoglycemia when patients fail to respond.

Primary Safety Endpoint:

The change in A1C from randomization to the end of the treatment period will be used to demonstrate that the automatic insulin delivery suspension (LGS ON) does not result in an unacceptable worsening of glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 16-21 years are determined by the investigator to have the appropriate, requisite support (family, caregiver or social network) to successfully participate in this study
* Subjects who are determined by the investigator to be psychologically sound in order to successfully participate in this study.
* Subject was < 40 years at disease onset
* Subject has been diagnosed with type 1 diabetes ≥ 2 years
* Subject is willing to perform ≥ 4 finger stick blood glucose measurements daily
* Subject is willing to perform required sensor calibrations
* Subject is willing to wear the system continuously throughout the study
* Subject is willing to keep a log to record at minimum:
* Sick days
* Days with exercise and days with symptoms of low glucose
* Subject has an A1C value 5.8% to 10.0% (as processed by Central Lab) at time of screening visit
* Subject must be on pump therapy use for >6 months prior to Screening
* Subject has been followed by a well trained diabetes health care provider(s) for 6 months prior to screening
* Subject is willing to upload data weekly from the study pump, must have Internet access and a computer system that meets the requirements for uploading the study pump
* If subject has celiac disease, it has been adequately treated as determined by the investigator
* Subject is willing to take one of the following insulins and can financially afford to use either of the 2 insulin preparations throughout the course of the study (i.e. co-payments for insulin with insurance or able to pay full amount)
* Humalog® (insulin lispro injection)
* NovoLog® (insulin aspart)

Exclusion Criteria:

* Subject has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening:
* Medical assistance (i.e. Paramedics, Emergency room or Hospitalization)
* Coma
* Seizures
* Subject is unable to tolerate tape adhesive in the area of sensor placement
* Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, rash, Staphylococcus infection)
* Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study
* Subject has had any of the following new diagnoses within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
* Subject is being treated for hyperthyroidism at time of screening
* Subject has an abnormality (out of upper reference range, as processed by Central Lab) in creatinine at time of screening visit
* Subject has an abnormality (out of reference range, as processed by Central Lab) in thyroid-stimulating hormone (TSH) at time of screening visit
* Subject has taken any oral, injectable, or IV steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study
* Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
* Subject has been hospitalized or has visited the emergency room in the 6 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes
* Subject is currently abusing illicit drugs
* Subject is currently abusing prescription drugs
* Subject is currently abusing alcohol
* Subject is using pramlintide (Symlin) at time of screening
* Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
* Subject has elective surgery planned that requires general anesthesia during the course of the study
* Subject is a shift worker with working hours between 10pm and 8am.
* Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
* Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
* Subject diagnosed with current eating disorder such as anorexia or bulimia
* Subject plans to use significant quantity of herbal preparations (use of over the counter herbal preparation for 30 consecutive days or longer period during the study) or significant quantity of vitamin supplements (four times the recommended daily allowance used for 30 consecutive days or longer period during the study) during the course of their participation in the study
* Subject has been diagnosed with chronic kidney disease that results in chronic anemia
* Subject is on dialysis

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Arkansas Diabetes Clinic and Research Center, Little Rock, Arkansas
  - AMCR Institute, Inc, Escondido, California
  - Frank Diabetes Research Institute/ Mills-Peninsula Health Center, San Mateo, California
  - University of Colorado Denver/ Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Metabolic Research Institute, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Physicians Research Associates, Lawrenceville, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountains Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Research Center, Des Moines, Iowa
  - International Diabetes Center, Minneapolis, Minnesota
  - Naomie Barrie Diabetes Center, New York, New York
  - Joslin Diabetes Center, Syracuse, New York
  - Ohio University College of Osteopathic Medicine, Athens, Ohio
  - Texas Diabetes, Austin, Texas
  - Rainier Clinical Research Center, Renton, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Weiss R, Garg SK, Bode BW, Bailey TS, Ahmann AJ, Schultz KA, Welsh JB, Shin JJ. Hypoglycemia Reduction and Changes in Hemoglobin A1c in the ASPIRE In-Home Study. Diabetes Technol Ther. 2015 Aug;17(8):542-7. doi: 10.1089/dia.2014.0306. Epub 2015 Jun 2. PMID 26237308
- [Derived] Weiss R, Garg SK, Bergenstal RM, Klonoff DC, Bode BW, Bailey TS, Thrasher J, Schwartz F, Welsh JB, Kaufman FR; ASPIRE In-Home Study Group. Predictors of Hypoglycemia in the ASPIRE In-Home Study and Effects of Automatic Suspension of Insulin Delivery. J Diabetes Sci Technol. 2015 May 18;9(5):1016-20. doi: 10.1177/1932296815586014. PMID 25986629
- [Derived] Klonoff DC, Bergenstal RM, Garg SK, Bode BW, Meredith M, Slover RH, Ahmann A, Welsh JB, Lee SW. ASPIRE In-Home: rationale, design, and methods of a study to evaluate the safety and efficacy of automatic insulin suspension for nocturnal hypoglycemia. J Diabetes Sci Technol. 2013 Jul 1;7(4):1005-10. doi: 10.1177/193229681300700424. PMID 23911183
- [Derived] Bergenstal RM, Klonoff DC, Garg SK, Bode BW, Meredith M, Slover RH, Ahmann AJ, Welsh JB, Lee SW, Kaufman FR; ASPIRE In-Home Study Group. Threshold-based insulin-pump interruption for reduction of hypoglycemia. N Engl J Med. 2013 Jul 18;369(3):224-32. doi: 10.1056/NEJMoa1303576. Epub 2013 Jun 22. PMID 23789889

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Glucose Suspend Feasure (LGS): According to randomization, Low Glucose Suspend (LGS) will be turned ON in the treatment arm of the study
  Medtronic MMT-754 Veo Insulin pump testing Low Glucose Suspend (LGS) feature : Automatic suspension of insulin delivery when glucose is low.
- Control Arm: The Low Glucose Suspend feature will not be available to subjects in the control arm
  Medtronic (NO LGS FEATURE ) using Paradigm® Revel™2.0 Pump : No Automatic suspension of insulin delivery when glucose is low.
Period: Overall Study
Arm/Group | Low Glucose Suspend Feasure (LGS) | Control Arm
Started | 121 | 126
Completed | 116 | 124
Not Completed | 5 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Device Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Glucose Suspend Feature (LGS): According to randomization, Low Glucose Suspend (LGS) will be turned ON in the treatment arm of the study
  Medtronic MMT-754 Veo Insulin pump testing Low Glucose Suspend (LGS) feature : Automatic suspension of insulin delivery when glucose is low.
- Total: Total of all reporting groups
Arm/Group | Low Glucose Suspend Feature (LGS) | Control Arm | Total
Number analyzed (Participants) | 121 | 126 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 110 | 114 | 224
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.83) | 44.8 (13.82) | 43.3 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 151
  Male | 46 | 50 | 96
Region of Enrollment [Number; unit: participants]
  United States | 121 | 126 | 247

OUTCOME MEASURES:

1. Primary Outcome: Change in A1C From Baseline to End of Study Participation
Description: The first study objective is to demonstrate that home use of Low Glucose Suspend (LGS) is safe and is not associated with glycemic deterioration, as measured by change in A1C from baseline to end of study participation.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Group A With Low Glucose Suspend (LGS) Feature Turned 'ON' | Group B Without Low Glucose Suspend (LGS) Feature
Number analyzed (Participants) | 116 | 124
Percent | 0.00 (0.44) | -0.04 (0.42)
Statistical Analysis 1: Comparison: Group A With Low Glucose Suspend (LGS) Feature Turned 'ON' vs Group B Without Low Glucose Suspend (LGS) Feature; Test type: Non-Inferiority or Equivalence — pre-specified non-inferiority margin of 0.4% was used for sample size calculation. sample size is based on two-sample t test with one-sided type 1 error of 2.5%. Assuming a same mean of change in A1C for the treatment arm and control arm and a common standard deviation of 1% for both treatment groups, it showed that a total of 200 subjects will provide over 80% power to detect the non-inferiority with a margin of 0.4%; ANCOVA; Mean Difference (Final Values) = 0.05, 97.5% CI 1-sided [upper limit 0.15]

2. Primary Outcome: The Event Area Under the Curve (AUC) Was Used to Demonstrate the Reduction of Nocturnal Hypoglycemia With the Low Glucose Suspend (LGS) Feature (LGS ON)
Description: An event is identified as: LGS feature in the correct setting; CGM values <= 65 mg/dL continuously with starting time between 10pm - 8am; No evidence of patient intervention during the first 20 minutes when CGM value was <= 65 mg/dL; The rate of change before reaching sensor glucose value of <= 65 mg/dL was <= 5 mg/dl/minutes; If the time between two successive events was less than 30 minutes, they will be combined as one event; An evaluable event is defined as any event with CGM value <= 65 mg/dL of greater than 20 minutes and the LGS feature is on the correct setting; Event AUC analysis was performed based on logarithm of AUC data.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: mg/dL x min
Arm/Group | Group A With Low Glucose Suspend (LGS) Feature Turned 'ON' | Group B Without Low Glucose Suspend (LGS) Feature
Number analyzed (Participants) | 121 | 126
mg/dL x min | 980 (1200.1) | 1568 (1994.9)
Statistical Analysis 1: Comparison: Group A With Low Glucose Suspend (LGS) Feature Turned 'ON' vs Group B Without Low Glucose Suspend (LGS) Feature; Test type: Superiority or Other; p < 0.025, ANCOVA; Mean Difference (Final Values) = -588

ADVERSE EVENTS:
Time Frame: Severe adverse event data and adverse event data were collected during approximately 4 months of study duration
Description: Adverse events during run-in (training) period are available upon request
Arm/Group | Group A With Low Glucose Suspend (LGS) Feature Turned 'ON' | Group B Without Low Glucose Suspend (LGS) Feature
Serious Adverse Events (participants affected / at risk) | 0/121 | 2/126
Other Adverse Events (participants affected / at risk) | 39/121 | 41/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A With Low Glucose Suspend (LGS) Feature Turned 'ON' (N=121) | Group B Without Low Glucose Suspend (LGS) Feature (N=126)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Not related to study device or study procedure
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Not related to study device or study procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A With Low Glucose Suspend (LGS) Feature Turned 'ON' (N=121) | Group B Without Low Glucose Suspend (LGS) Feature (N=126)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomit (Gastrointestinal disorders) | 1 (1) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1)
Dental bridge failure (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Application site bleeding (General disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis Acute (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Infusion Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Track Infection (Infections and infestations) | 3 (4) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Vaginal Mycosis (Infections and infestations) | 2 (2) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1)
Stomach Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No